CLINICAL TRIAL: NCT02518828
Title: High Versus Low SpO2 Oxygen Therapy in Patients With Acute Heart Failure
Acronym: HiLo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other); Alberta Innovates Health Solutions (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HiLo-HF- 2 Pilot Trial
Record Dates: First submitted 2015-08-04; First posted 2015-08-10 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2017-11

CONDITIONS: Heart Failure
Keywords: Acute Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (2):
- High SpO2 (Active Comparator): In the high SpO2 set-point arm, patients will have a nasal cannula placed and will be manually titrated to SpO2 range ≥96%
  Interventions: Other: High SpO2
- Low SpO2 (Active Comparator): In the low SpO2 set-point arm, patients will have a nasal cannula placed and will be manually titrated to SpO2 range 90-92%
  Interventions: Other: Low SpO2

INTERVENTIONS:
Other: High SpO2 — SpO2 range ≥96%
  Arms: High SpO2
Other: Low SpO2 — SpO2 range 90-92%
  Arms: Low SpO2

SUMMARY:
The primary objective of this pilot trial is to determine whether inpatients presenting to the Emergency Department (ED) with symptoms suggestive of Acute Heart Failure (AHF), who receive supplemental oxygen adjusted at either a high (SpO2 range ≥96%) or low (SpO2 range 90-92%) oxygen saturation level, leads to greater reduction in N-terminal-proBNP (NT-proBNP) at 72 hours.

DETAILED DESCRIPTION:
Patients will be randomized to either a high (SpO2 range ≥96%) or low (SpO2 range 90-92%) oxygen after informed consent.

ELIGIBILITY:
Inclusion Criteria:

* >40 years of age presenting to the ED with AHF
* objective finding of HF (BNP >400 pg/ml or Chest X-Ray with pulmonary congestion)
* plan to admit with primary diagnosis as HF
* must be able to be randomized within 16 hours of presenting to the ED
* provided written informed consent

Exclusion Criteria:

* on home oxygen
* known prior hypercapnic failure (PaCO2 >50 mmHg)
* asthma
* primary pulmonary hypertension,
* patients who require urgent positive pressure ventilation or intubation
* patients on >10 L/min oxygen

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Change in NT-proBNP from baseline to 72 hours | 72 hours

SECONDARY OUTCOMES:
Change in dyspnea using the visual analog scale (VAS) from baseline to 72 hours | 72 hours
Change in global symptoms using the Patient Global Assessment scale (PGA) from baseline to 72 hours | 72 hours
Change in Peak Expiratory Flow Rate (PEFR) from baseline to 72 hours | 72 hours
Number of worsening heart failure (WHF) events | 7 days
30-day clinical events | 30 days
  All cause mortality, HF readmission, days alive and out of hospital
Average z-score from the combination of these outcomes: PGA, NT-proBNP, 7-day WHF, 30-day mortality and re-hospitalization | 30 days
Hochberg endpoint (combination of NT-proBNP and PGA) | 72 hours
Diuretic response (weight loss up to 72 hours and urine volume up to 24 hours) | 72 hours

OTHER OUTCOMES:
Safety Outcome - Need for mechanical ventilation (invasive and non-invasive | 7 days
  Number of participants with post-enrollment respiratory failure with a need for mechanical ventilation as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Justin Ezekowitz, MBBCH, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital / Mazankowski Alberta Heart Institute, Edmonton, Alberta, Canada